CLINICAL TRIAL: NCT05198505
Title: Phase I Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of TQB2868 Injection in Subjects With Advanced Malignant Tumors
Brief Title: Clinical Trial of TQB2868 Injection in Subjects With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2868-I-01
Record Dates: First submitted 2022-01-19; First posted 2022-01-20 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2868 Injection (Experimental): The drug was administered once every 3 weeks (administration time window: ± 3 days), the dose of each administration was 1.5-600 mg, and 3 weeks was a treatment cycle until the disease progressed or the investigator judged that it was not suitable to continue the drug use.
  Interventions: Drug: TQB2868 Injection

INTERVENTIONS:
Drug: TQB2868 Injection — TQB2868 protein is a bi-functional fusion protein targeting PD-1 and TGF-β

SUMMARY:
The TQB2868 protein in this study targeted programmed cell death protein 1 (PD-1) and transforming growth factor-β (TGF-β). The bifunctional fusion protein targets and neutralizes TGF-β in the tumor microenvironment. On the basis of inhibiting PD-1 / programmed death ligand 1 (PD-L1) pathway, T cells can restore activity, enhance immune response, and more effectively improve the effect of inhibiting tumor occurrence and development.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects voluntarily join the study and sign an informed consent form.
* 2 Age: 18-75 years old (when signing the informed consent form); Eastern Cooperative Oncology Group Performance status (ECOG PS) score: 0~1 points.
* 3 Advanced malignant tumors clearly diagnosed by histology or cytology.
* 4 Patients with advanced malignant tumors who have been diagnosed by tissue and/or cytology and have failed standard treatments or lack effective treatment options.
* 5 The main organs are in good function, and the following examination results are good: routine blood examination, biochemical examination, blood coagulation function examination, heart color Doppler ultrasound evaluation.
* 6 Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study; serum pregnancy/urine within 7 days before study entry The pregnancy test is negative and must be a non-lactating subject; male subjects should agree that contraception must be used during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* 1 Combined diseases and medical history:

  1. Has had other malignant tumors within 3 years before the first medication. The following two conditions can be included in the group: other malignant tumors treated with a single operation to achieve disease-free survival (DFS) for 5 consecutive years; cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [ Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  2. Unrelieved toxic reactions higher than Common Terminology Criteria Adverse Events (CTC AE) level 1 or higher caused by any previous treatment, excluding hair loss;
  3. Major surgical treatment, obvious traumatic injury or long-term unhealed wounds or fractures have been received within 28 days before the first medication;
  4. Arterial/venous thrombosis occurred within 6 months before the first administration, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
  5. Existence of active pulmonary tuberculosis, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment or active pneumonia with clinical symptoms;
  6. People who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
  7. Previous recipients of allogeneic bone marrow transplantation or solid organ transplantation.
  8. Subjects with any severe and / or uncontrolled disease.
* 2 Tumor-related symptoms and treatment:

  1. Have received chemotherapy, radiotherapy or other anti-cancer therapies within 4 weeks before the first medication (the washout period will be calculated from the end of the last treatment); if you have received local radiotherapy in the past, you can join the group if the following conditions are met: End of radiotherapy more than 4 weeks from the start of the study treatment (brain radiotherapy is more than 2 weeks); and the target lesion selected for this study is not in the radiotherapy area; or the target lesion is located in the radiotherapy area, but progress has been confirmed.
  2. Received Chinese patent medicine treatment with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions within 2 weeks before the first medication;
  3. Have previously received immunological double-antibody therapeutic drugs against the same target of TQB2868 injection;
  4. Uncontrollable pleural effusion, pericardial effusion or ascites that still needs to be drained repeatedly (investigator's judgment);
  5. Known to have spinal cord compression, cancerous meningitis, accompanied by brain metastasis symptoms, or symptom control time less than 2 weeks;
* 3 Research and treatment related:

  1. The history of live attenuated vaccine vaccination within 28 days before the first administration or the planned live attenuated vaccine vaccination during the research period;
  2. Those who have had severe hypersensitivity reactions after using macromolecular drugs;
  3. An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, corticosteroids, or immunosuppressive agents) occurred within 2 years before the first medication. Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
  4. Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose>10mg/day prednisone or other curative hormones), and continue within 2 weeks of the first administration in use;
* 4 Participated in other anti-tumor drug clinical trials within 4 weeks before the first medication;
* 5 According to the judgment of the researcher, there are situations that seriously endanger the safety of the subjects or affect the completion of the research by the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | up to 10 months
  DLT definition: the subject has the following adverse events related to the test drug within one treatment cycle (21 days) after the first administration.
  1. Grade ≥ 3 neutropenia with fever; Grade 4 neutropenia that cannot be recovered within 3 days after symptomatic treatment; Grade 3 anemia that cannot be recovered within 14 days;
     ≥ Grade 3 thrombocytopenia with bleeding; Other hematological toxicity above grade 4 (inclusive);
  2. ≥ Grade 3 non hematological toxicity; Nausea, vomiting, diarrhea, rash and electrolyte disorder that cannot be recovered to grade ≤ 2 within 7 days after symptomatic treatment; Grade 3 general fatigue, fatigue and headache with duration ≥ 7 days; Laboratory examination abnormalities with isolated ≥ grade 3 and significant clinical symptoms;
  3. Adverse events related to ≥ grade 3 infusion reaction occurred, and did not return to normal within 6 hours after stopping infusion
Recommended Phase II Dose (RP2D) | up to 10 months
  To evaluate RP2D of TQB2868 injection in adult patients with advanced malignant tumors
Maximum Tolerated Dose (MTD) | up to 10 months
  Defined as the highest dose when dose-limiting toxicity (DLT) occurred in less than 33% of subjects.
All adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs) | up to 17 months
  ncidence of all adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs)

SECONDARY OUTCOMES:
Time to reach maximum(peak )plasma concentration following drug administration (Tmax) | up to 17 months
  To characterize the pharmacokinetics of TQB2868 by assessment of time to reach maximum plasma concentration after single and multiple dosing
Maximum (peak) plasma drug concentration (Cmax) | up to 17months
  Cmax is the maximum plasma concentration of TQB2868.
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Css-max) | up to 17 months
  Cmax is the steady state maximum concentration of TQB2868 .
Title：The plasma concentration time curve at steady state, from 0 to τ area under curve of time. (AUC0-τ) | up to 17 months
  To characterize the pharmacokinetics of TQB2868 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | up to 17 months
  To characterize the pharmacokinetics of TQB2868 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Area under the plasma concentration-time curve from time zero to infinity(AUC0-∞) | up to 17 months
  To characterize the pharmacokinetics of TQB2868 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Apparent total clearance of the drug from plasma after oral administration (CL/F) | up to 17 months
  CL/F is total clearance rate for TQB2868.
Elimination half-life (t1/2) | up to 17 months
  t1/2 is time it takes for the blood concentration of TQB2868 to drop by half.
Apparent volume of distribution of intravenous infusion(Vss/F) | up to 17 months
  Steady-state apparent volume of distribution of TQB2868 injection by intravenous infusion
Elimination rate constant(λ) | up to 17 months
  λ is the elimination rate constant when TQB2868 participates in the calculation of metabolism in the body
Area under the plasma concentration-time curve from time zero to time 24h.( AUC0-24h) | up to 17 months
  Characterize the pharmacokinetics of TQB2868 by evaluating the area under the plasma concentration-time curve from the first administration to 24h
Mean residence time (MRT) | up to 17 months
  MRT describes the average time that TQB2868 remains in the body.
Minimum steady-state plasma drug concentration during a dosage interval (Css-min) | up to 17 months
  Css-min is the minimum plasma concentration of TQB2868.
Degree of fluctuation(DF) | up to 17 months
  DF is the volatility coefficient of TQB2868.
Average steady-state plasma drug concentration during multiple-dose administration (Css-avg) | up to 17 months
  Css-avg is the average of steady-state plasma concentration of TQB2868 .
Anti-drug antibodies(ADA) | up to 17 months
  ADA is antibodies that make TQB2868 clear in the body quickly
Receptor Occupancy(RO) | up to 17 months
  RO is a receptor occupancy for TQB2868 involved in metabolism in the body
Progression-free survival (PFS) | up to 29 months
  PFS is defined as the time from the first treatment to the first disease progression or death from any cause
Overall response rate (ORR) | up to 29 months
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 29 months
  Percentage of participants achieving CR and PR and stable disease (SD).
Duration of Response (DOR) | up to 29 months
  The period from the participants first achieving CR or PR to disease progression.
Overall survival (OS) | up to 29 months
  OS is defined as the time from the first administration to all-cause death.
PD-L1 expression in tumor tissue | up to 17 months
  To evaluate the expression of PD -L1
TGF-β expression in blood samples | up to 17 months
  To evaluate the expression of TGF-β

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality